CLINICAL TRIAL: NCT05847296
Title: The Second Affiliated Hospital of Nanchang University
Brief Title: Effect of Preoperative Sarcopenia on Postoperative Delirium in Elderly Patients Undergoing Gastrointestinal Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Principal Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Other Study IDs: 2023-OB-01
Record Dates: First submitted 2023-04-13; First posted 2023-05-06 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Postoperative Delirium; Sarcopenia; Gastrointestinal Surgery; Anesthesia
Keywords: Postoperative Delirium; Sarcopenia; Gastrointestinal surgery; Anesthesia
MeSH Terms: conditions — Emergence Delirium; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Sarcopenia group
- Non sarcopenic group

SUMMARY:
The goal of this observational study is to compare Incidence of postoperative delirium in Sarcopenic and non-sarcopenic elderly patients undergoing gastrointestinal surgery. The main question it aims to answer are:

• Effect of preoperative sarcopenia on postoperative delirium in elderly patients undergoing gastrointestinal surgery Participants will be evaluated preoperatively for sarcopenia and assessed for postoperative delirium, pain, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 65 years old, gender is not limited
2. Patients to undergo elective abdominal surgery (gastrointestinal tumor resection) under general anesthesia, with an expected operation duration of about 2h~4h
3. ASA Ⅰ-Ⅲ

Exclusion Criteria:

1. Relative contraindications to general anesthesia: Patients with severe heart and lung disease, severe infection, uncontrolled hypertension, diabetes, and severe diabetic complications
2. Abnormal renal and liver function: AST or ALT≥2.5×ULN, TBIL≥1.5×ULN, Serum creatinine concentration (SCC)≥1.5×ULN
3. People with a history of mental illness or long-term use of psychotropic drugs (dementia, schizophrenia), chronic analgesic drug use, alcoholism, and cognitive impairment
4. Any cardiovascular or cerebrovascular accidents occurred within 3 months, such as myocardial infarction, stroke, transient ischemic attack
5. Myasthenia gravis patients
6. Unable to cooperate to complete the test, the patient or family member rejected the participant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All patients who come to the Second Affiliated Hospital of Nanchang University for treatment
Sampling Method: Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative delirium | Within 7 days after surgery. Delirium at any time during the 7 days after surgery was considered postoperative delirium.
  Postoperative delirium was assessed using the 3D-CAM scale. It consists of 4 features, and a positive feature 1 and 2 plus 3 or 4 is considered postoperative delirium.

SECONDARY OUTCOMES:
Systolic pressure | Up to 5 hours in the operating room
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Diastolic pressure | Up to 5 hours in the operating room
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Mean pressure | Up to 5 hours in the operating room
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Heart rate | Up to 5 hours in the operating room
  "just entering the operating room", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the operating room".
Incidence of postoperative admission to ICU | Up to 1 month after surgery
  Including immediate postoperative admission to ICU and postoperative admission to ICU in the ward.
Length of stay in ICU | Up to 1 month after surgery
  Duration of stay in ICU after surgery
Postoperative pain | Within 7 days after surgery
  The degree of postoperative pain was assessed using the Numerical Rating Scale (NRS). The pain level increased sequentially from 0-10
Maximum postoperative C-reactive protein (CRP) | Up to 1 month after surgery
  Only the highest CRP values detected in the normal course of gastrointestinal surgery are collected, and no additional blood sampling or interventions are performed
Minimum postoperative albumin | Up to 1 month after surgery
  Only the lowest albumin values detected in the normal course of gastrointestinal surgery are collected, and no additional blood sampling or interventions are performed
Length of hospitalization | After the patient is discharged from the hospital, average 1 month
  The total number of days the patient spent at the hospital for the current consultation
Complication | During the perioperative period, up to 1 month after surgery
  All the perioperative complications are recorded

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital of Nanchang University, Nanchang University, Nanchang, Jiangxi, China